CLINICAL TRIAL: NCT04264286
Title: The Effects of Esmolol on the Hemodynamic Response to Orotracheal Extubation: a Prospective, Randomized, Double-blind and Placebo-controlled Trial
Brief Title: The Effects of Esmolol on the Hemodynamic Response to Orotracheal Extubation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, Preceptor of Medical Residency in Anesthesiology, Hospital de Base
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Esmolol and extubation
Record Dates: First submitted 2020-02-05; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Beta Blocker; Hemodynamic Instability
Keywords: Esmolol; Extubation; Hemodynamic instability

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind and placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esmolol group (Active Comparator): Patients will receive intravenous esmolol after the end of the surgical procedure.
  Interventions: Drug: Prophylactic esmolol
- Placebo group (Placebo Comparator): Patients will receive intravenous saline after the end of the surgical procedure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prophylactic esmolol — Patients will receive prophylactic esmolol after the end of the surgery
  Arms: Esmolol group
Drug: Placebo — Patients will prophylactic placebo after the end of the surgery
  Arms: Placebo group

SUMMARY:
Beta-blockers are useful tools for the prevention of hemodynamic instability in the manipulation of airways. The main objective of the present study is to evaluate the effectiveness of using esmolol in attenuating hemodynamic responses at the time of tracheal extubation, by assessing the incidence of tachycardia in relation to placebo.

DETAILED DESCRIPTION:
The moment of extubation represents a critical period of anesthesia where important hemodynamic changes occur. These occur due to stimulation of the larynx, trachea and bronchi that generates an increased release of catecholamines. In high-risk patients, these hemodynamic changes can have serious consequences.

Many strategies have been used to control the hemodynamic response to airway manipulation during the period of intubation, but until today there is no standard therapy for this control during the period of extubation. Therefore, the investigators aim to study the use of beta-blockers in this context.

Beta-blockers are an attractive pharmacological strategy as they reduce the activation of the sympathetic nervous system proper at this time. Esmolol, due to its short half-life, can be an ideal tool to ensure better hemodynamic control.

There are few studies in the literature that study this drug during extubation, and there is no consensus on the best dose or method of administration for this moment.

Therefore, this study aims to evaluate the effectiveness of using esmolol in attenuating hemodynamic responses at the time of tracheal extubation, by assessing the incidence of tachycardia in relation to placebo.

This prospective, randomized, double-blind, placebo-controlled study aims to verify the hypothesis that esmolol reduces hemodynamic instability induced by tracheal extubation in surgical procedures at Base Hospital of the Federal District. The examiners responsible for patient assessment will not have access to the agents used.

Patients will be randomized through a randomly generated list. The examiner responsible for opening the envelope will make the draw, will include the patient in one of the groups, write down their data in the random list, prepare the syringe with the medication, and deliver it to the operating room so that the next examiners will not be aware of the administered drug.

Patients will receive standard general anesthesia and after the end of the surgical procedure, patients will be allocated the study drug (esmolol 2 mg/kg) or placebo group. All patients will receive sugammadex as a reversal of neuromuscular block and monitored appropriately.

The evolution of vital signs such as systolic blood pressure, mean heart rate, incidence and intensity of adverse events such as cough, bucking, bradycardia, tachycardia, hypertension, hypotension, vasopressor and anticholinergic consumption will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 60 years, electively scaled for surgery requiring general anesthesia.
* Physical State 1, 2 or 3 of the American Society of Anesthesiology (ASA)

Exclusion Criteria:

* Patients with cardiac disease
* Patients with renal disease
* Patients with liver disease
* Patient with lung disease
* Patients using beta blockers or calcium channel blockers
* Patients who refuse to participate in the study after presenting the informed consent form

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as tachycardia | Through study completion, an average of 15 minutes (during awakening from anesthesia)
  Intraoperative hemodynamic stability analysis through the incidence tachycardia

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio T Mendonça, MD, MSc, Principal Investigator — Hospital de Base do Distrito Federal
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Federal District, Brazil